CLINICAL TRIAL: NCT02417870
Title: Safety and Efficacy of Treatment With Ultra-low Dose Subcutaneous IL-2 to Promote Regulatory T Cells Post Renal Transplantation
Brief Title: Ultra-low Dose Subcutaneous IL-2 in Renal Transplantation
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of funding/resources
Sponsor: Anil K. Chandraker, MD (Other)
Responsible Party: Sponsor-Investigator, Anil K. Chandraker, MD, Medical Director of Kidney and Pancreas Transplantation, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015P000796
Record Dates: First submitted 2015-04-13; First posted 2015-04-16 (Estimated); Results first posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Kidney Transplantation
Keywords: Transplantation; interleukin-2; IL-2; Kidney; Renal
MeSH Terms: interventions — aldesleukin; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- aldesleukin (Experimental)
  Interventions: Biological: aldesleukin

INTERVENTIONS:
Biological: aldesleukin
  Other Names: recombinant IL-2; recombinant interleukin-2; proleukin

SUMMARY:
To investigate the safety and tolerability of treatment with low dose rIL-2 in renal transplant recipients. To assess the immunologic impact of low dose rIL-2 in renal transplant recipients. To assess the efficacy of low dose rIL-2 in renal transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients
* >18 years and <75 years of age
* >6 months post Tx
* on stable dose of immunosuppression
* Transplant biopsy showing interstitial fibrosis and tubular atrophy of grade II or greater, with some evidence of lymphocytic infiltration (biopsy is NOT a study procedure, it would be performed as part of the patient's SOC)
* Ability to give informed consent

Exclusion Criteria:

* Biopsy proven acute cellular rejection; greater than grade 1A
* Baseline creatinine >3.5mg/dL
* Patients with active infection, including Hepatitis B and C, HIV
* Current or prior invasive malignancy
* Patients who are pregnant or breastfeeding
* Patients who are unable to give consent
* Prior intolerance of/allergy to IL2
* Inability to comply with treatment
* History of thrombotic angiopathy including hemolytic uremic syndrome and thrombotic thrombocytopenic purpura
* Symptomatic congestive cardiac failure or uncontrolled cardiac angina
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
* WOCBP and male subjects with reproductive potential must agree to use a highly effective method of birth control [defined in protocol & ICF] during study treatment, and for 6 months after completion of treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Anil Chandraker, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Aldesleukin: aldesleukin
Period: Overall Study
Arm/Group | Aldesleukin
Started | 2
Completed | 0
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Aldesleukin
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Increase in Treg Count
Time Frame: 6 weeks
Population: Study was termination prior to completion
Arm/Group | Aldesleukin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Aldesleukin
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aldesleukin (N=2)
ischemic heart disease (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aldesleukin (N=2)
Elevated Creatinine (General disorders) | 2 — associated with advanced kidney disease and other comorbidities

LIMITATIONS AND CAVEATS:
Both enrolled subjects were discontinued prior to completion due to adverse events associated with advanced kidney disease and other comorbidities. The study was closed to enrollment in 2017 and ultimately terminated prior to completion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-09): https://cdn.clinicaltrials.gov/large-docs/70/NCT02417870/Prot_SAP_000.pdf